CLINICAL TRIAL: NCT02519829
Title: A Randomized Clinical Trial Comparing Monocryl and Dermabond Closure Versus Staple Closure in Total Hip Arthroplasty
Brief Title: A Clinical Trial Comparing Monocryl and Dermabond Closure Versus Staple Closure in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, James Howard, Assistant Professor, Orthopedic Surgery, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6757 (REB # 16747)
Record Dates: First submitted 2015-05-28; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Unilateral Primary Osteoarthritis, Unspecified Hip
Keywords: Suture; Skin staples; Vicryl; Monocryl
MeSH Terms: interventions — Polyglactin 910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monocryl closure (Active Comparator): The skin incision is closed with monocryl dissolvable sutures and a topical adhesive (glue) called Dermabond and covered with a Tegaderm dressing.
  Intervention: Monocryl closure, Tegaderm dressing
  Interventions: Procedure: Monocryl closure; Procedure: Tegaderm dressing
- Vicryl and staple closure (Active Comparator): The skin incision is closed with vicryl and staples and covered with a gauze dressing.
  Intervention: Vicryl and Staple closure, Gauze dressing
  Interventions: Procedure: Vicryl and Staple closure; Procedure: Gauze dressing

INTERVENTIONS:
Procedure: Monocryl closure — Total Hip Arthroplasty with monocryl closure of wound
  Arms: Monocryl closure
Procedure: Vicryl and Staple closure — Total Hip Arthroplasty with vicryl and staple closure of wound
  Arms: Vicryl and staple closure
Procedure: Tegaderm dressing — Total Hip Arthroplasty with monocryl closure of wound and tegaderm dressing
  Arms: Monocryl closure
Procedure: Gauze dressing — Total Hip Arthroplasty with vicryl and staple closure of wound and gauze dressing
  Arms: Vicryl and staple closure

SUMMARY:
Patients undergoing primary hip arthroplasty will be randomized to receive either monocryl closure of fascial and dermal layers with dermabond and tegaderm covering versus standard vicryl closure of fascia layer and staple closure for skin. Short term wound complications, pain and patient and surgeon-rated cosmetic scar appearance will be measured. The investigators will also measure operating room time and costs associated with dressing changes and wound-related procedures (e.g. staple removal).

DETAILED DESCRIPTION:
Wound closure has always been based on surgeon preference and type of closure. Skin closure is considered the most important part of the surgical procedure by some since it is often the only visible evidence of the surgical procedure. In fact, conclusions about the success of the surgery are often based on the appearance of the wound.

There have been a few studies in a variety of surgical journals that have looked at the two pertinent methods of closure with the majority coming from obstetrical journals comparing caesarian section closure with staples versus a subcuticular monocryl suture. For the most part, although patient satisfaction is quite high initially for a subcuticular closure, at long term follow-up patient satisfaction scores are quite similar.

One study published in the Journal of Bone and Joint Surgery recommended that staple closure was more beneficial for skin closure than monocryl sutures for total hip and knee arthroplasty. Their recommendations were based on an overall shorter operative time when using staple closure compared to monocryl sutures. They also found that final patient satisfaction and complication rates were relatively similar 3 months postoperatively. This group published an earlier paper as well describing the use of glue for closure and did report an decrease in overall drainage rates when they analyzed their data for subcuticular sutures as opposed to staples.

A more recent study evaluated wound appearance at 3 months using a surgeon -rated visual analogue scale to compared the use of adhesive tapes versus staples for skin closure following total hip arthroplasty. Again, no significant difference in patient satisfaction scores were reported.

To date, there is a paucity of well-powered studies to compare outcomes in patients whose wounds are closed using the usual staple methods compared to a monocryl suture method. In addition, outcomes have focused on surgeon-ratings and not patient ratings. The proposal for this study is to compare overall patient and surgeon-rated cosmetic scar appearance and complications following total hip replacement with skin closure for using monocryl suture versus staples. This study would use a more recent, validated assessment tool than the VAS scale. The assessment is called the Patient Observer Scar Assessment Scale (POSAS ) and it incorporates six essential features about the wound such as colour, malleability, etc. The form is split so that the surgeon rating carries the same weight in the final score as the patient assessment of their own scar. This scale gives a nice balance for determining overall satisfaction and wound healing combining surgeon and patient scores.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 100 years old
2. Undergoing total hip replacement

Exclusion Criteria:

1. Previous scar over newly planned incision
2. Alcoholism
3. Mentally unfit to complete questionnaire
4. Connective tissue disease and/or psoriasis/eczema/dermatitis
5. Previous joint infection at surgical site
6. Any use of immunosuppressive medications or disease modifying agents
7. Medical contra-indication to surgery
8. Pregnancy
9. Lack of permanent home address
10. Drug Abuse
11. Allergy to Skin Adhesive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient Observer Scar Assessment Scale for overall patient satisfaction rates. | 3 months
  Questionnaire

SECONDARY OUTCOMES:
Wound complications | 2 week, 6 week, 3 month post-operatively
  Analysis - number of participants with wound complications
Drainage rates | 2 week, 6 week, 3 month post-operatively
  Analysis - number of participants with wound drainage
Need for post-operative antibiotics | 2 week, 6 week, 3 month post-operatively
  Analysis - number of participants with need for post-operative antibiotics
Patient pain score | 2 week, 6 week, 3 month post-operatively
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: James L Howard, MD, Principal Investigator — London Health Sciences Centre